CLINICAL TRIAL: NCT02331095
Title: A Pilot Study of Using Statins in Patients With Acute Venous Thromboembolism (VTE)
Brief Title: Statin Use in Patients With Acute VTE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Tzu-Fei Wang, Associate professor of Internal Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014H0262
Record Dates: First submitted 2014-12-22; First posted 2015-01-06 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Atorvastatin; Anticoagulation Bridge; Warfarin; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anticoagulation (Active Comparator): Patients will be treated with warfarin with dose adjusted to goal International Normalized Ratio (INR) of 2-3 or rivaroxaban standard dose (15 mg twice daily for 3 weeks then 20 mg daily)
  Interventions: Drug: Anticoagulation Therapy
- Atorvastatin + anticoagulation (Experimental): In addition to standard anticoagulation, patients will be given concurrent atorvastatin 40 mg daily for the study period of 9 months, starting from the time of enrollment
  Interventions: Drug: Atorvastatin; Drug: Anticoagulation Therapy

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin belongs to the "statin" class of drugs, and is routinely used for prevention of cardiovascular diseases and/or reduction of cholesterol levels. It has been shown to decrease the risk of first venous thromboembolism in an otherwise healthy population with elevated high-sensitivity C-reactive protein (hs-CRP).
  Other Names: Lipitor
  Arms: Atorvastatin + anticoagulation
Drug: Anticoagulation Therapy — Warfarin is a standard anticoagulation in the treatment for venous thromboembolism. The dose will be adjusted to goal INR of 2-3.
  Other Names: warfarin or rivaroxaban

SUMMARY:
This is a pilot, randomized, open-labelled study. Eligible patients will be enrolled and randomized 1:1 into "anticoagulation" arm or "anticoagulation plus atorvastatin" arm, with atorvastatin given at 40 mg orally daily for 3 months. The targeted total accrual is 80 patients, with 40 in each arm. Patients will be recruited from the hospitals and clinics at The Ohio State University Wexner Medical Center. Follow up visits are planned at enrollment, 3 months, and 9 months after randomization. At each follow up, blood will be obtained and assessments will include structured interviews of signs and symptoms of recurrent venous thromboembolism (VTE), bleeding, post thrombotic syndrome, and adverse events from study drugs.

DETAILED DESCRIPTION:
VTE is a potentially life-threatening disease, with an estimated incidence of 1-2 per 1000. Despite anticoagulation as standard of care, many patients still suffer from its complications: 30% will have VTE recurrence after an unprovoked VTE, and 25-50% will develop post-thrombotic syndrome. Therefore, there is an urgent need for effective therapies to reduce long-term VTE morbidities. Limitations in our understanding of the underlying pathophysiology of VTE and the absence of accurate biomarkers are significant problems. Without this knowledge, improvement in treatment is unlikely. Therefore, the overall objective of the study is to determine important biomarker changes in acute VTE and the actions of innovative adjunct therapy on those biomarkers. The rationale of the study is that, once the biomarker changes following acute VTE and the actions of therapies are established, treatment for acute VTE could be improved.

Statins are effective in the prevention of arterial thrombosis. Recently, arterial and venous thromboses are shown to share common pathophysiological mechanisms, and effective therapies for arterial thrombosis could provide benefits in VTE. Several observational studies and the JUPITER trial, a large, randomized, placebo-controlled study, have demonstrated that statins significantly reduce the risk of first VTE by 40%. Additionally, as few as 3 days of atorvastatin increase plasma fibrin clot permeability and susceptibility to lysis. Statins have been commonly prescribed for many other medical conditions such as coronary artery diseases and hyperlipidemia, and have demonstrated good safety profiles. These promising results, as well as their safety profiles, make statins an attractive potential addition to the standard anticoagulation for treating acute VTE, in an effort to reduce long-term morbidity. The effects of statins on thrombin generation in patients with acute VTE have not been studied. A study in patients with atrial fibrillation on warfarin showed a 40% reduction in endogenous thrombin potential with only three months of intensive cholesterol-lowering treatment including statins. Similar effects could be seen in patients with acute VTE. In addition, previous studies evaluating the effects of statins on the reduction of D-dimer or inflammatory cytokines revealed promising results but were not focused on patients with acute VTE. Therefore, this study will generate important information for acute VTE patients. This is a pilot, randomized, open-labelled study. Eligible patients will be enrolled and randomized 1:1 into "anticoagulation" arm or "anticoagulation plus atorvastatin" arm, with atorvastatin given at 40 mg orally daily for 3 months. The targeted total accrual is 80 patients, with 40 in each arm. Patients will be recruited from the hospitals and clinics at The Ohio State University Wexner Medical Center. Follow up visits are planned at enrollment, 3 months, and 9 months after randomization. At each follow up, blood will be obtained and assessments will include structured interviews of signs and symptoms of recurrent venous thromboembolism (VTE), bleeding, post thrombotic syndrome, and adverse events from study drugs. The primary objective of the study is to determine the reduction of thrombin peak concentration and/or endogenous thrombin potential measured by Thrombin Generation Assay (TGA) at 3 months in the "anticoagulation +atorvastatin" arm as compared to the "anticoagulation" arm. The secondary objectives are to determine the chronological changes of hemostatic, inflammatory, and lipidomic biomarker profiles in patients with acute VTE receiving anticoagulation as standard of care, with and without statins. The biomarker profile of interest, in addition to thrombin generation, include: D-dimer, Interleukin- 6 (IL-6), Interleukin-8 (IL-8), tumor necrosis factor (TNF)-α, high sensitivity C-reactive protein, free fatty acids, lipoprotein-associated phospholipase A2 , pro- inflammatory eicosanoids. The ultimate goal is to study the mechanisms of VTE and use of statin in VTE patients. Other secondary objectives include determination of relevant clinical outcomes such as VTE recurrence, VTE related mortality, arterial thrombosis, hemorrhage, post thrombotic syndrome, and residual vein obstruction in patients receiving standard of care versus standard of care plus statins.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* A diagnosis of proximal DVT (proximal to and including popliteal vein), with or without PE, confirmed by objective imaging studies, such as Doppler ultrasound, venograms (for DVT) and/or computer tomography, angiograms, ventilation-perfusion scan (for PE)
* Treated with warfarin as anticoagulation (short-term bridging with heparin or lovenox is allowed)

Exclusion Criteria:

* Thrombolysis within 6 weeks prior to enrollment
* Patients with statin use within 6 weeks of enrollment
* Patients with known allergy or intolerance to statins or statins are contraindicated for any other reasons
* Patients with baseline aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin ≥2.0 x upper limit of normal (ULN)
* Pregnant or breastfeeding females are excluded
* Any malignancy diagnosed within the preceding 2 years, except for squamous cell carcinoma or basal cell carcinoma of skin treated with local resection only, or carcinoma in situ of the cervix
* Incarcerated patients are excluded from the study due to the inherent difficulties in maintaining close follow-up for study purposes in patients who are incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10-27 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Fei Wang, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Wang TF, Waller AP, Lin E, Wei L, Bartosic A, Riedl K, Kerlin BA. A pilot randomized trial of atorvastatin as adjunct therapy in patients with acute venous thromboembolism. Blood Coagul Fibrinolysis. 2021 Jan 1;32(1):16-22. doi: 10.1097/MBC.0000000000000968. PMID 33196511

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin + Anticoagulation: In addition to warfarin or rivaroxaban as standard anticoagulation, patients will be given concurrent atorvastatin 40 mg daily for 3 months, starting from the time of enrollment
  Atorvastatin: Atorvastatin belongs to the "statin" class of drugs, and is routinely used for prevention of cardiovascular diseases and/or reduction of cholesterol levels. It has been shown to decrease the risk of first venous thromboembolism in an otherwise healthy population with elevated high-sensitivity C-reactive protein (hs-CRP).
  Warfarin: Warfarin is a standard anticoagulation in the treatment for venous thromboembolism. The dose will be adjusted to goal INR of 2-3.
  Atorvastatin: Atorvastatin belongs to the "statin" class of drugs, and is routinely used for prevention of cardiovascular diseases and/or reduction of cholesterol levels. It has been shown to decrease the risk of first venous thromboembolism in an otherwise healthy population with elevated high-sensitivity C-reactive protein (hs-CRP).
Period: Overall Study
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Started | 11 | 10
Completed | 7 | 9
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 54 [22 to 63] | 57.5 [48 to 72] | 55 [22 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 8 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasions | 10 | 7 | 17
  African Americans | 1 | 3 | 4
Pulmonary Embolism (PE) (in addition to DVT) [Count of Participants; unit: Participants] | 2 | 2 | 4
Provoked [Count of Participants; unit: Participants] — A provoked VTE is one with no identifiable provoking event; such as: surgery, malignancy, major trauma, significant immobility, pregnancy, or hormone therapy within 3 months prior to the event.
  Participants | 8 | 6 | 14
Hemoglobin (g/dL) [Median (Full Range); unit: g/dL] | 13.7 [10.3 to 16] | 12.1 [9.4 to 15.5] | 13.4 [9.4 to 16]
Platelet count (K/uL) [Median (Full Range); unit: K/uL] | 276 [194 to 664] | 301 [165 to 608] | 290 [165 to 664]
Creatinine (mg/dL) [Median (Full Range); unit: mg/dL] | 0.82 [0.52 to 1.34] | 0.74 [0.4 to 0.91] | 0.77 [0.4 to 1.34]

OUTCOME MEASURES:

1. Primary Outcome: The Reduction of Endogenous Thrombin Potential
Description: Determine the reduction of endogenous thrombin potential measured by Thrombin Generation Assay (TGA) at 3 months in the "anticoagulation +atorvastatin" arm as compared to the "anticoagulation" arm.
Time Frame: 3 Months
Measure: Median (Full Range); unit: nM*min
Groups:
- Atorvastatin + Anticoagulation: In addition to warfarin or rivaroxaban as standard anticoagulation, patients will be given concurrent atorvastatin 40 mg daily for 3 months, starting from the time of enrollment
  Atorvastatin: Atorvastatin belongs to the "statin" class of drugs, and is routinely used for prevention of cardiovascular diseases and/or reduction of cholesterol levels. It has been shown to decrease the risk of first venous thromboembolism in an otherwise healthy population with elevated high-sensitivity C-reactive protein (hs-CRP).
  Warfarin: Warfarin is a standard anticoagulation in the treatment for venous thromboembolism. The dose will be adjusted to goal INR of 2-3.
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
nM*min
  Enrollment | 1155 [0 to 1853] | 1440 [0 to 3190]
  3 Months | 1275 [0 to 2562] | 1143 [60 to 3766]

2. Primary Outcome: The Reduction of Peak Thrombin Concentration
Description: Determine the reduction of thrombin peak concentration measured by Thrombin Generation Assay (TGA) at 3 months in the "anticoagulation +atorvastatin" arm as compared to the "anticoagulation" arm.
Time Frame: 3 Months
Measure: Median (Full Range); unit: nM
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
nM
  Enrollment | 37 [0 to 157] | 67 [0 to 123]
  3 Months | 54 [0 to 149] | 48 [11 to 253]

3. Secondary Outcome: The Composite Rate of Recurrent Venous Thromboembolism (VTE) and VTE Related Mortality
Description: Recurrent PE was defined as new filling defect(s) seen on CT angiogram or a new high-probability ventilation-perfusion lung scan (22, 23). Recurrent DVT was defined as new uncompressible segments seen on vascular Doppler ultrasonography in a previously uninvolved limb, clearly extending from the prior thrombosis, or a new venous segment in a previously involved limb.
Time Frame: 3 months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
Participants
  3 Months | 0 | 0
  9 Months | 0 | 0

4. Secondary Outcome: The Rate of Arterial Thrombotic Events
Description: Arterial thromboembolism was defined a new myocardial infarction (based on typical electrocardiographic findings and/or elevation of cardiac enzymes) or cerebral vascular accident (based on clinical syndrome of development of focal or global loss of brain function thought to be vascular in origin, confirmed by appropriate standard imaging studies).
Time Frame: 3 months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
Participants
  3 Months | 0 | 0
  9 Months | 0 | 0

5. Secondary Outcome: The Rate of Residual (Chronic) Vein Obstruction by Doppler Ultrasound
Description: Residual venous obstruction was assed by Doppler Ultrasonography. Residual chronic DVT (to any degree) was reported.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
Participants | 8 | 8

6. Secondary Outcome: The Reduction of Clinical Post-thrombotic Syndrome (PTS), as Objectively Evaluated With Villalta Scoring System
Description: The Villata score for Post-Thrombotic Syndrome (PTS) stratifies the severity of post-thrombotic syndrome in lower extremity DVT. The score contains a combination of 5 subjective symptoms as reported by the patient (cramps, itching, pins and needles, heaviness, and pain) and 6 objective signs measured by a provider (edema, skin induration, hyperpigmentation, prominent veins on legs, redness, and tenderness on calf compression). Each sign is scaled from 0 (no or minimal) to 3 (severe) with a total score ranged from 0 to 33. Higher scores represent more severe disease.
Time Frame: 3 Months
Measure: Median (Full Range); unit: scores on a scale
Groups:
- Anticoagulation: Patients will be treated with warfarin as standard anticoagulation, dose adjusted to goal International Normalized Ratio (INR) of 2-3
  Warfarin: Warfarin is a standard anticoagulation in the treatment for venous thromboembolism. The dose will be adjusted to goal INR of 2-3.
- Atorvastatin + Anticoagulation: In addition to warfarin as standard anticoagulation, patients will be given concurrent atorvastatin 40 mg daily for 3 months, starting from the time of enrollment
  Atorvastatin: Atorvastatin belongs to the "statin" class of drugs, and is routinely used for prevention of cardiovascular diseases and/or reduction of cholesterol levels. It has been shown to decrease the risk of first venous thromboembolism in an otherwise healthy population with elevated high-sensitivity C-reactive protein (hs-CRP).
  Warfarin: Warfarin is a standard anticoagulation in the treatment for venous thromboembolism. The dose will be adjusted to goal INR of 2-3.
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
scores on a scale
  Enrollment | 7 [0 to 18] | 4.5 [2 to 21]
  3 Months | 6 [1 to 13] | 3.5 [0 to 15]

7. Secondary Outcome: The Rate of Major, Non-major, and All Hemorrhages Defined by the International Society on Thrombosis and Haemostasis (ISTH) Criteria
Description: Major bleeding events were defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria, with overt bleeding in critical organs (e.g. central nervous system, retroperitoneum), a >2 gram/dL drop in hemoglobin from baseline, or requiring at least two units of packed red blood cell transfusion meeting the criteria for major bleeding. Clinically relevant, non-major bleeding (CRNMB) events were defined as any other bleeding events reported by patients but not otherwise meeting the above listed criteria for major bleeding.
Time Frame: 3 months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
Participants
  3 Months | 0 | 0
  9 Months | 0 | 0

8. Secondary Outcome: Change in the Levels of D-Dimer at 3 Months
Time Frame: 3 Months
Measure: Median (Full Range); unit: mcg/mL FEU
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
mcg/mL FEU
  Enrollment | 2.12 [0.88 to 13.78] | 2.2 [0.6 to 5.42]
  3 Months | 0.36 [0.27 to 0.71] | 0.59 [0.27 to 1.23]

9. Secondary Outcome: Change in the Levels of C-Reactive Protein at 3 Months
Description: C-Reactive (CRP) was measured using high sensitivity.
Time Frame: 3 Months
Measure: Median (Full Range); unit: mg/L
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
mg/L
  Enrollment | 5.5 [2 to 51.4] | 7.0 [2 to 42.4]
  3 Months | 3.9 [0.6 to 15.7] | 5.1 [0.9 to 21.1]

10. Secondary Outcome: Change in Low-Density Lipoproteins (LDL) at 3 Months
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
mg/dL
  Enrollment | 123.8 (22.73) | 116.9 (43.07)
  3 Months | 115.9 (30.63) | 76.1 (26.02)

11. Secondary Outcome: Change in Triglyceride Levels at 3 Months
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
Number analyzed (Participants) | 11 | 10
mg/dL
  Enrollment | 130.5 (47.69) | 157.9 (83.06)
  3 Months | 127.4 (60.45) | 135.3 (83.79)

ADVERSE EVENTS:
Time Frame: At each visit (enrollment, 3 and 9 months), patients will be evaluated by physicians and study personnel for any adverse events and any side effects from statins and/or anticoagulation.
Arm/Group | Anticoagulation | Atorvastatin + Anticoagulation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Our study was limited by the small sample size, early termination due to low recruitment rate and lack of funding. The protocol was amended to include patients on rivaroxaban (initially only warfarin). Lost to follow up is also significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02331095/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02331095/ICF_001.pdf